CLINICAL TRIAL: NCT05720845
Title: Effects of Different Ventilatory Strategy on Intraoperative Atelectasis During Bronchoscopy Under General Anesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of Department of Respiratory Medicine, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20230111
Record Dates: First submitted 2023-01-12; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Lung Disorder
Keywords: atelectasis; general anesthesia
MeSH Terms: conditions — Lung Diseases; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional mechanical ventilation (Active Comparator): Conventional mechanical ventilation for General Anesthesia
  Interventions: Procedure: conventional mechanical ventilation
- VESPA (Experimental): ventilatory strategy to prevent atelectasis for General Anesthesia
  Interventions: Procedure: VESPA

INTERVENTIONS:
Procedure: VESPA — Using Ventilatory strategy of prevent atelectasis for General Anesthesia.
  Arms: VESPA
Procedure: conventional mechanical ventilation — Conventional mechanical ventilation for General Anesthesia.
  Arms: conventional mechanical ventilation

SUMMARY:
This trial compares two different types of ventilation for the prevention of partial or complete collapsed lung (atelectasis) in patients undergoing interventional pulmonology procedures under general anesthesia. Ventilatory strategy to prevent reduce the intra-procedural development of atelectasis during interventional pulmonology procedures under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing interventional pulmonology procedures with radial probe endobronchial ultrasound (RP-EBUS) for peripheral lung lesions
* Recent (< 4 weeks) chest computed tomography (CT) performed prior to the bronchoscopy

Exclusion Criteria:

* Patients with baseline lung consolidation, interstitial changes or lung masses (> 3 cm in diameter) in dependent areas of the lung (right/left [R/L] B6, 9, or 10 bronchial segments) as seen on most recent CT
* History of primary or secondary spontaneous pneumothorax

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-08 (Estimated); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-03-18 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of new atelectasis for each segment | During bronchoscopy, an average of 1 hour.
  The proportion of patients identified as developing intraprocedural atelectasis by radial probe endobronchial ultrasound (RP-EBUS)

SECONDARY OUTCOMES:
Ventilation-induced complications | Within 48 hours of bronchoscopy
Bronchoscopy-induced complications | Within 48 hours of bronchoscopy
Assess the regional ventilation distribution by Electrical impedance tomography (EIT) | During bronchoscopy, an average of 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China